CLINICAL TRIAL: NCT01106105
Title: Impact of Obesity on Postural Control
Status: Completed | Type: Observational
Sponsor: Université Joseph Fourier (Other)
Other Study IDs: PCO
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2010-04

CONDITIONS: Balance; Postural Control; Mechanical Factor

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control (Body Mass Index < 25)
- Obese (Body Mass Index > 35)

SUMMARY:
The goal of the present study was to objectively evaluate the postural behaviour of type II obese patients as compared to adults showing a normal body mass index (BMI) in critical postural tasks.

ELIGIBILITY:
Inclusion:

* BMI > 35 or BMI < 25

Exclusion:

* Muscular, neurological or cardiovascular deficits
* Competitive physical activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ten healthy non-obese adults (control group, age = 42.4 ± 15.1, BMI = 22.4 ± 1.3, five women and five men) and ten obese adults (obese group, age = 46.2 ± 19.6, BMI = 35.2 ± 2.8, five women and five men, F(1,18)=0.3, p>0.05, and F(1,18)=176.3, p<.001, for control vs. obese age and BMI, respectively) voluntarily took part in this investigation.
Sampling Method: Non-Probability Sample
Dates: Start 2010-04